CLINICAL TRIAL: NCT02934711
Title: Establish a Quality Rating Scale for Primary Care Centers and Nursing Homes Pluri Professionals Integrating the Perspective of Patients in Complex Situations and Their Caregivers
Brief Title: A Quality Rating Scale for Patients in Complex Situations and Their Caregivers
Acronym: QualSoPrim
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC16.0144
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2019-04

CONDITIONS: Patients in Complex Situations
Keywords: Multimorbidity; Exercise coordinated groups (GECO); Caregivers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Identify and analyze in the exercise groups coordinated (GECO) the effects of coordination arrangements between professionals on the transformation of modes of exercise of professional care, and on the experience of patients / users and that of caregivers, particularly on dimensions constituted that the quality of care in order to build a coordinated exercise structures rating scale primary care on the basis of criteria suggested by patients

ELIGIBILITY:
Inclusion Criteria:

* For Professionals:
* Medical or paramedical professionals working in the exercise coordinated groups (GECO) initially defined
* Professionals who made his non_opposition
* For patients and family caregivers:
* Binomials patients / caregivers over the age of 18.
* Binomials patients / caregivers who formulated his non_opposition
* Patients experiencing complex care (multi-morbid and chronic)

Exclusion Criteria:

* Refusal of a participant (Professionals / Patients / caregivers) to respond to inquiries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In each of exercise coordinated groups (GECO), it will be important to obtain a variety of cases studied in terms of socio-demographic characteristics (although populations of the basins of different exercise coordinated groups may have more or less specific profiles, to be taken into account) and range previous care.
  The population of multimorbid patients and caregivers will be vary with regard to age, sex, place of residence (living alone or cohabiting with relatives or hosted) and professional categories
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2018-01-24 (Actual)

PRIMARY OUTCOMES:
A quality assessment scale | 18 months
  Perform a quality assessment scale for primary care in the exercise coordinated groups (GECO) of perspective in complex situations patients, their caregivers and healthcare professionals

CONTACTS AND LOCATIONS:
Locations (1):
- Maison de santé de l'Aulne Maritime du Faou, Le Faou, France, France

IPD SHARING:
Plan to Share IPD: No